CLINICAL TRIAL: NCT00541359
Title: A Phase I Trial of PS-341 in Combination With Topotecan in Advanced Solid Tumor Malignancies
Brief Title: Bortezomib and Topotecan Hydrochloride in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03109; NCI-2009-01598 (Registry Identifier: NCI CTRP); CDR0000570257 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib; Topotecan; trioctyl phosphine oxide; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): PART I (completed as of 09/06/06; all patients enrolled in study after 09/06/06 are enrolled in part II): Patients receive escalating doses of topotecan hydrochloride IV over 30 minutes on days 1 and 8 followed 6 hours later by bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.
  PART II: Patients receive bortezomib IV on days 1, 4, 8, and 11 followed 6 hours later by escalating doses of topotecan hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.
  In both parts of the study, patients who achieve a response may receive additional courses of treatment.
  Interventions: Drug: bortezomib; Drug: topotecan hydrochloride; Other: immunohistochemistry staining method; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with topotecan hydrochloride may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of topotecan hydrochloride when given together with bortezomib in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of combining PS-341 with topotecan in patients with advanced solid tumor malignancies.

II. To define the maximum tolerated dose (MTD) of topotecan when administered in combination with a fixed dose of PS-341 and to described the toxicities at each dose studied.

III. To evaluate the pharmacokinetics of topotecan when given in combination with PS-341 at MTD.

SECONDARY OBJECTIVES:

I. To perform laboratory correlative studies on patients tissue investigating potential predictors of response.

OUTLINE:

PART I (completed as of 09/06/06; all patients enrolled in study after 09/06/06 are enrolled in part II): Patients receive escalating doses of topotecan hydrochloride IV over 30 minutes on days 1 and 8 followed 6 hours later by bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.

PART II: Patients receive bortezomib IV on days 1, 4, 8, and 11 followed 6 hours later by escalating doses of topotecan hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.

In both parts of the study, patients who achieve a response may receive additional courses of treatment.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* Histologic proof of solid tumor malignancy
* ANC >= 1500/microliter
* PLT >= 150,000/microliter
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* AST =< 2.5 x ULN or AST =< 5 x ULN if liver involvement
* Serum creatinine =< 1.5
* Life expectancy >= 12 weeks
* ECOG performance status 0, 1, or 2
* Subjects with asymptomatic brain metastases are allowed

Exclusion

* ECOG PS 3 or 4
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have received chemotherapy or radiation therapy for at least four weeks, and they must have recovered from any toxicities of previous treatment (ongoing grade 1 dermatologic toxicities are allowable)
* Eligible patients should not be taking enzyme-inducing anticonvulsants due to the potential of pharmacokinetic interactions
* Pregnant and nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD] or abstinence, etc.)
* Other concurrent chemotherapy, immunotherapy, or radiotherapy
* HIV-positive patients receiving anti-retroviral therapy (HAART); there is a potential for pharmacokinetic interactions
* Bisphosphonate therapy (e.g. pamidronate or zoledronate) will not be considered investigational agents for the purpose of trial eligibility
* Pre-existing grade >= 2 neuropathy
* No previous treatment with PS-341 allowed, however there is no limit to other prior therapy with chemotherapy, including topotecan, and radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0 | 21 days after the end of treatment

SECONDARY OUTCOMES:
Overall survival | 1 year from the end of treatment
Progression-free survival | 1 year from the end of treatment
Time to progression | 1 year from the end of treatment
Levels of NF-kB activation | At baseline and completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Cristea, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Medical Group Inc, Pasadena, California